CLINICAL TRIAL: NCT00531024
Title: Systemic Bevacizumab (Avastin) Therapy for Exudative Neovascular Age-Related Macular Degeneration
Brief Title: Systemic Avastin Therapy in Age-Related Macular Degeneration
Acronym: BEAT-AMD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Prof.Dr. Susanne Binder M.D., Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-043-0505
Record Dates: First submitted 2007-09-15; First posted 2007-09-18 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Macular Degeneration
Keywords: Exudative Neovascular; AMD; Avastin; Systemic; Exudative Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 3 intravenous infusions of 5mg/kg bevacizumab at 2 weeks intervals
  Interventions: Drug: Bevacizumab
- 2 (Placebo Comparator): 3 intravenous infusions of 100ml sodium chloride 0,9% at 2 weeks intervals
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Bevacizumab — 3 intravenous infusions of 5mg/kg bevacizumab at 2 weeks intervals
  Other Names: Avastin
  Arms: 1
Drug: Sodium Chloride — 3 intravenous infusions of 100ml sodium chloride 0,9% at 2 weeks intervals
  Arms: 2

SUMMARY:
Choroidal neovascularisation (CNV) in age-related macular degeneration is one of the major causes of blindness in the western world. It is already known that the vascular endothelial growth factor (VEGF) plays a major role in the development of CNV. Photodynamic therapy (PDT), subretinal surgery, and intravitreal injection of VEGF- inhibitors are the common treatments. These methods are either very invasive or need to be repeated several times over long periods of time in order show some effect. Furthermore PDT can only be performed in eyes with pigment epithelium detachments (PED) of maximum 50% of the avascular zone, while intravitreal injections can lead to endophthalmitis and acute glaucoma. A systemic treatment, which would only need to be administered 3 times within 6 weeks would be a major effort in macular degeneration therapy.

DETAILED DESCRIPTION:
Bevacizumab (Avastin®, Genentech Inc.) is a new anti-vascular endothelial growth factor (anti-VEGF) which has shown promising results as a combination therapy with 5-fluorouracil, leucovorin, and oxaliplatin in first-line treatment of metastatic colorectal cancer14,15. Since intraocular anti-VEGF therapies for CNV in AMD have already shown promising results, the idea of this study is to administer the anti-VEGF bevacizumab intravenously, as a systemic therapy, in AMD-patients.

The rationale of the present study is to determine the effect of systemic bevacizumab therapy in patients with fibrovascular pigment epithelium detachment (PED), involving the geometric center of the foveal avascular zone, in comparison to placebo treatment with sodium chloride 0,9%.

The patients will receive 3 intravenous infusions of 5mg/kg bevacizumab at 2 weeks intervals or 3 intravenous infusions of 100ml sodium chloride 0,9% at 2 weeks intervals. Medical internal reviews, ETDRS and Radner visual acuity assessment, ophthalmologic examinations, ocular imaging with OCT 3, multifocal ERG, fluorescein angiography, and indocyanine angiography will be performed. The follow-up time is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* AMD patients with fibrovascular pigment epithelium detachment (PED), subfoveal choroidal neovascularisations (CNV) extending under the geometric center of the foveal avascular zone, and a central retinal thickness of at least 300 microns.

Exclusion Criteria:

* Patients who had arterial thromboembolic diseases
* Patients with: Cancer, Proteinuria, Renal impairment, Hepatic dysfunction, Vision threatening ophthalmic diseases other than AMD

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Lesion size | 6 months

SECONDARY OUTCOMES:
Macular thickness, visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Katharina E Schmid-Kubista, MD, Study Director — LBI
Locations (1):
- Dept. of Ophthalmology, Rudolf Foundation Clinic, Vienna, Vienna, Austria